CLINICAL TRIAL: NCT03466281
Title: Structured Patient Group Education Versus Structured Patient Education Via the Internet for Patients With Irritable Bowel Syndrome (IBS)
Brief Title: Patient Education for Patients With Irritable Bowel Syndrome (IBS)
Acronym: IBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Magnus Simrén, Professor, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IBS patient education
Record Dates: First submitted 2017-11-29; First posted 2018-03-15 (Actual); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Patient Education; IBS - Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: Active Comparator: 1 Structured patients group intervention - IBS School Active Comparator: 2 Structured Patient education via Internet
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IBS School (Active Comparator): Patient education provided in a group setting
  Interventions: Behavioral: Structured patient group education
- Internet patient education (Active Comparator): Patient education provided via the internet
  Interventions: Behavioral: Education via Internet

INTERVENTIONS:
Behavioral: Structured patient group education — Patient education in a group setting
  Arms: IBS School
Behavioral: Education via Internet — Patient education via the internet
  Arms: Internet patient education

SUMMARY:
In this randomized controlled study in patients with irritable bowel syndrome (IBS) the investigators plan to compare the effects of a structured patient group education (IBS School) with structured education provided via the internet. The effects of the interventions on GI and psychological symptom severity, knowledge and quality of life will be assessed with validated questionnaires at baseline, immediately after the intervention and 3 and 6 months after the intervention.

DETAILED DESCRIPTION:
In this randomized controlled study in patients with irritable bowel syndrome (IBS) the investigators plan to compare the effects of a structured patient group education (IBS School), which previously has been evaluated and found to efficacious for symptom improvement (1-3), with a similar education provided via the internet in a non-inferiority design. The investigators hypothesize that structured patient education provided via the internet is not inferior compared to structured patient group education.

Men and women from 18 years of age, with IBS according to the Rome III criteria, who are referred from physicians in primary care and secondary/tertiary care to receive patient education will be included. The education, both the IBS School and the internet based version, will be managed at the GI outpatient clinic at Sahlgrenska University hospital in Gothenburg. Patients with an organic GI disease and/or with another disease potentially affecting the GI symptoms are excluded. Likewise, patients with a disability to communicate in the Swedish language or to use a computer and/or do not have access to a computer or internet are excluded.

Moreover, patients with a severe psychiatric disease are excluded due to potential problems to participate in a group intervention. In order to allocate an equal number of patients to both of the interventions during the study, a number of up to 20 patients will be invited in a block and the patients will be randomly divided into two groups with an equal number of patients in each group. The groups will then be randomized 1:1 to either start the IBS School or to start the patient education via internet within two to three weeks. After the randomization all patients will receive a personal login to the database and an e-mail with information on how to log in and complete the questionnaires online. All questionnaires will be completed by the patients on-line, i.e. all data will be registered directly into the database.

The interventions:

Both interventions in the study are designed based on the self-efficacy theory, and the general theory of nursing. Moreover, the education is performed based on a biopsychosocial model considered to be important in functional GI disorders. The IBS School consists of three, two hour sessions held once per week in a group setting with eight to ten patients in each group. A nurse and a dietician lead the education and issues are chosen with the aim to cover a wide spectrum of issues related to IBS. A lot of space is given for discussion within the group. At the first session, general information is provided about IBS, symptoms, pathophysiology and treatment options. At the second session, food related issues is discussed and at the third session the effects from other life style factors like stress, physical activity and relaxation is discussed.

The patient education provided via the internet covers the same areas of issues related to IBS that are covered in the structured group education. The participants in the internet group will receive and read information which is divided into three steps, once weekly. At the end of each treatment week the patients will have a contact via the internet with the nurse and dietician and thereby receive feedback on questions that were raised during the treatment week. The patients are also encouraged to attend (anonymously) a specific, closed internet forum where they have the opportunity to discuss and reflect over information material from the last week with other patients attending the internet based intervention. The time consumed to read the information and reflect is estimated to two hours weekly.

ELIGIBILITY:
Inclusion Criteria:

* IBS according to the Rome III criteria

Exclusion Criteria:

* organic GI disease and/or another disease potentially affecting the GI symptoms
* severe psychiatric disease due to potential problems to participate in a group intervention
* disability to communicate in the Swedish language
* disability to use a computer or not have access to a computer or internet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-11-20 (Actual)

PRIMARY OUTCOMES:
Change of GI symptoms | Measuring change from Baseline and up to six months after the education
  Measured with a questionnaire; Irritable Bowel Syndrome-severity scoring system (IBS-SSS). Five issues measure the severity of IBS symptoms on a scale, each ranging from 0 to 100. A total score is calculated ranging from 0 to 500. In this study the total score is used, the higher the score the worse severity of symptoms.

SECONDARY OUTCOMES:
Change of Quality of life | Measuring change from Baseline and up to six months after the education
  Measured with a questionnaires; Irritable Bowel Syndrome Quality Of Life (IBSQOL) is a disease-specific HRQOL instrument, including 30 items measuring nine dimensions of health, emotional functioning, mental health, sleep, energy, physical functioning, diet, social role, physical role and sexual relations. Raw scores are transformed into a scale of 0-100, with 100 representing the best possible quality of life scores for each of the nine dimensions.
Change of Psychological symptoms | Measuring change from Baseline and up to six months after the education
  Measured with a questionnaire; Hospital Anxiety and Depression scale (HAD). This scale consists of 14 items with seven items relating to anxiety and seven to depression. A four-graded scale was used (0-3), giving a total range from 0 to 21 on each subscale. The higher the score, the more pronounced the symptom. HAD was developed for nonpsychiatric medical patients to detect anxiety and depression.
Change of GI specific anxiety | Measuring change from Baseline and up to six months after the education
  Measured with a questionnaire; Visceral Sensitivity Index (VSI) which is a 15-item (each question ranging from 0 to 5) questionnaire designed to measure the degree of GI-specific anxiety in IBS. The total score ranges from 0 (no GI-specific anxiety) to 75 (severe GI-specific anxiety), and the higher the score, the higher the GI-specific anxiety
Change of Perceived knowledge about IBS | Measuring change from Baseline and up to six months after the education
  Measured with a Visual Analogue scale (VAS). The patients were asked to rate their perceived knowledge of IBS on a Visual Analog Scale (VAS). The scale comprised a 100-mm straight line with the extremes labeled 'No knowledge at all' and 'Very much knowledge'. The score ranges from 0 to 100 and the higher the score the more perceived knowledge of IBS.

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Simren, MD, Prof, Principal Investigator — Dept of internal medicine, Gothenburg University
Locations (1):
- Dept of Internal Medicine, Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ringstrom G, Storsrud S, Lundqvist S, Westman B, Simren M. Development of an educational intervention for patients with Irritable Bowel Syndrome (IBS): a pilot study. BMC Gastroenterol. 2009 Feb 4;9:10. doi: 10.1186/1471-230X-9-10. PMID 19192312
- [Result] Ringstrom G, Storsrud S, Posserud I, Lundqvist S, Westman B, Simren M. Structured patient education is superior to written information in the management of patients with irritable bowel syndrome: a randomized controlled study. Eur J Gastroenterol Hepatol. 2010 Apr;22(4):420-8. doi: 10.1097/MEG.0b013e3283333b61. PMID 19923998
- [Result] Ringstrom G, Storsrud S, Simren M. A comparison of a short nurse-based and a long multidisciplinary version of structured patient education in irritable bowel syndrome. Eur J Gastroenterol Hepatol. 2012 Aug;24(8):950-7. doi: 10.1097/MEG.0b013e328354f41f. PMID 22617366
- [Derived] Lindfors P, Axelsson E, Engstrand K, Storsrud S, Jerlstad P, Tornblom H, Ljotsson B, Simren M, Ringstrom G. Online Education Is Non-Inferior to Group Education for Irritable Bowel Syndrome: A Randomized Trial and Patient Preference Trial. Clin Gastroenterol Hepatol. 2021 Apr;19(4):743-751.e1. doi: 10.1016/j.cgh.2020.04.005. Epub 2020 Apr 11. PMID 32289541